CLINICAL TRIAL: NCT02034552
Title: A Randomized Open-label Phase IIa Study Evaluating Quantified Bone Scan Response Following Treatment With Radium-223 Dichloride Alone or in Combination With Abiraterone Acetate or Enzalutamide in Subjects With Castration-resistant Prostate Cancer Who Have Bone Metastases
Brief Title: A Randomized Phase IIa Efficacy and Safety Study of Radium-223 Dichloride With Abiraterone Acetate or Enzalutamide in Metastatic Castration-resistant Prostate Cancer (CRPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16544
Record Dates: First submitted 2013-12-16; First posted 2014-01-13 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride; Abiraterone Acetate; Prednisone; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (3):
- Radium-223 dichloride (Xofigo, BAY88-8223) (Experimental)
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)
- Radium-223 with abiraterone&prednisone (Experimental)
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223); Drug: Abiraterone acetate; Drug: Prednisone
- Radium-223 with enzalutamide (Experimental)
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223); Drug: Enzalutamide

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Radium-223 dichloride (Xofigo, BAY88-8223) 50 kBq/kg (55 kBq/kg after implementation of NIST [National Institute of Standards and Technology] update) every 4 weeks x 6 doses intravenous slow bolus
Drug: Abiraterone acetate — Abiraterone acetate 1000 mg (4 x 250 mg tablets) taken orally once daily for up to two years following last dose of radium-223 dichloride
  Arms: Radium-223 with abiraterone&prednisone
Drug: Prednisone — Prednisone 5 mg capsule taken orally twice daily for up to two years following last dose of radium-223 dichloride
  Arms: Radium-223 with abiraterone&prednisone
Drug: Enzalutamide — Enzalutamide 160 mg (four 40 mg capsules) taken orally once daily for up to two years following last dose of radium-223 dichloride
  Arms: Radium-223 with enzalutamide

SUMMARY:
The primary objective in this study is to evaluate bone scan response at Week 24 based on the quantified technetium-99 bone scan lesion area (BSLA). The safety of radium-223 dichloride in combination with abiraterone acetate or enzalutamide will be investigated. The study will evaluate radiological progression free survival, overall survival, and skeletal events. This study will also explore the clinical utility of different imaging modalities (whole body quantified technetium-99 bone scan, DW-MRI [diffusion-weighted magnetic resonance imaging] and NaF [sodium fluoride] PET-CT [positron emission tomography-computed tomography] scan) and will have a separate central radiological review for applicable secondary and exploratory imaging endpoints. All subjects will be randomized as assigned randomly by the IXRS (interactive voice / web response system) system in a 1:1:1 ratio into one of the treatment arms: radium-223 dichloride alone, 50 kBq/kg (55 kBq/kg after implementation of NIST [National Institute of Standards and Technology] update) every 4 weeks for up to 6 doses; radium-223 dichloride, 50 kBq/kg (55 kBq/kg after implementation of NIST update) every 4 weeks up to 6 doses together with abiraterone acetate 1,000 mg daily and prednisone 5 mg bid (twice daily); radium-223 dichloride 50 kBq/kg (55 kBq/kg after implementation of NIST update) every 4 weeks up to 6 doses together with enzalutamide 160 mg daily. The study will consist of screening, treatment and follow-up periods. Study will continue until disease progression as determined by investigator, or when patient meets criteria for withdrawal from study. Subjects in treatment arms with abiraterone/prednisone or enzalutamide will have the option to continue taking oral study therapy until the end of the study (2 years from the last dose of radium-223 dichloride) if the investigator deems the subject may benefit and there is no clinical or radiological progression. Subjects who discontinue all study treatment prior to 2 years from last radium-223 dichloride treatment will enter active follow-up. During the active follow-up period, the subject will have a safety visit at the clinic every 12 weeks from the EOT (end of treatment) for up to 2 years from the last dose of radium-223 dichloride. Beyond 2 years from last radium-223 dichloride treatment,subjects will enter long-term follow-up and will be followed via phone contact at intervals to assess for safety (hematological toxicity and new primary malignancies) and overall survival. A separate long-term safety follow-up study protocol is planned. Once implemented, the study subjects surviving after the end of the active follow-up will be transitioned to this separate long-term safety follow-up protocol.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Known castration-resistant disease
* Serum PSA ≥2 ng/mL (μg/L)
* Multiple skeletal metastases (≥2 hot spots) on bone scan
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 2.
* Life expectancy ≥6 months
* Adequate hematologic, hepatic, and renal function

Exclusion Criteria:

* History of visceral metastasis, or visceral metastases
* Malignant lymphadenopathy with lymph nodes exceeding 3 cm in short axis diameter
* Medical condition that would make prednisone (corticosteroid) use contraindicated
* Any chronic medical condition requiring a higher dose of corticosteroid than 5 mg prednisone bid
* Treatment with more than one chemotherapy agent for prostate cancer
* Prior systemic radiotherapy and hemibody external radiotherapy
* History of pituitary or adrenal dysfunction
* Chronic conditions associated with non-malignant abnormal bone growth (e.g., confirmed Paget's disease of bone)
* Atrial fibrillation, or other cardiac arrhythmia requiring medical therapy
* History of seizures (taking/not taking anticonvulsants), arteriovenous malformation in the brain, head trauma with loss of consciousness
* Central nervous system (CNS) metastases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-03-07 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2018-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (19):
- United States (19):
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Los Angeles, California
  - New Haven, Connecticut
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Plantation, Florida
  - Indianapolis, Indiana
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Rockville, Maryland
  - Detroit, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - Syracuse, New York
  - The Bronx, New York
  - Springfield, Oregon
  - Houston, Texas
  - Seattle, Washington

REFERENCES:
- [Derived] Petrylak DP, Vaishampayan UN, Patel KR, Higano CS, Albany C, Dawson NA, Mehlhaff BA, Quinn DI, Nordquist LT, Wagner VJ, Siegel J, Trandafir L, Sartor O. A randomized phase IIa study of quantified bone scan response in patients with metastatic castration-resistant prostate cancer (mCRPC) treated with radium-223 dichloride alone or in combination with abiraterone acetate/prednisone or enzalutamide. ESMO Open. 2021 Apr;6(2):100082. doi: 10.1016/j.esmoop.2021.100082. Epub 2021 Mar 19. PMID 33744812

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 19 study centers in USA from 7-Mar-2014 (first subject's first visit) to 26-Jun-2018 (last subject's last visit).
Pre-assignment Details: Overall, 103 subjects were screened. Of them, 68 subjects were randomized, and 63 subjects were received study treatment.
Groups:
- Radium-223 Dichloride (Xofigo, BAY88-8223): Participants received radium-223 dichloride 50 kBq/kg (55 kBq/kg after implementation of National Institute of Standards and Technology (NIST) update) every 4 weeks x 6 doses IV (slow bolus).
- Radium-223 With Abiraterone & Prednision: Participants received radium-223 dichloride 50 kBq/kg (55 kBq/kg after implementation of NIST update) every 4 weeks x 6 doses (IV slow bolus), abiraterone acetate 1000 mg daily, and prednisone 5 mg bid (oral). The first dose of oral co-medications is to be given after the first radium-223 dichloride injection.
- Radium-223 With Enzalutamide: Participants received radium-223 dichloride 50 kBq/kg (55 kBq/kg after implementation of NIST update) every 4 weeks x 6 doses (IV slow bolus) and enzalutamide 160 mg daily (oral). The first dose of oral co-medications is to be given after the first radium-223 dichloride injection.
Period: Overall Study
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Radium-223 With Abiraterone & Prednision | Radium-223 With Enzalutamide
Started | 22 | 24 | 22
Received Treatment | 19 | 22 | 22
Completed | 8 | 4 | 5
Not Completed | 14 | 20 | 17
Not completed — Never treated | 3 | 2 | 0
Not completed — Radiological progression | 3 | 5 | 4
Not completed — AE not assoc. with disease progression | 1 | 4 | 2
Not completed — AE associated with disease progression | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Non-compliance with study drug | 0 | 0 | 1
Not completed — Clinical progression | 5 | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Radium-223 With Abiraterone & Prednision | Radium-223 With Enzalutamide | Total
Number analyzed (Participants) | 22 | 24 | 22 | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.5 (10.2) | 68.6 (8.6) | 71.0 (8.7) | 70.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 22 | 24 | 22 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 21 | 23 | 20 | 64
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 5 | 3 | 10
  White | 18 | 17 | 17 | 52
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 3
Eastern Cooperative Oncology Group [Count of Participants; unit: Participants] — ECOG = Eastern cooperative oncology group PS levels are 0 (Fully active, able to carry on all pre-disease performance), 1 (ambulatory and able to carry out work of a light or sedentary), 2 (Ambulatory and capable of all selfcare but unable to carry out any work activities), 3 (Capable of only limited selfcare, confined to bed or chair more than 50% of awake time), 4 (Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair) and 5 (death).
  Participants
    Missing | 3 | 2 | 0 | 5
    PS 0 | 10 | 13 | 11 | 34
    PS1 | 9 | 9 | 11 | 29

OUTCOME MEASURES:

1. Primary Outcome: Patient Bone Scan Response Rate
Description: Radiological bone scan response based on change from baseline of digitized technetium-99 bone scans using computer-aided detection software. Responder (R): 30% or greater resolution of the BSLA compared to baseline. Stable Disease (SD): Not meeting the criteria for R, PD, or UE. Progressive Disease (PD): Two or more new areas of radiotracer uptake attributable to metastatic disease in regions of bone that had not previously shown radiotracer uptake or greater than 30% increase from baseline in BSLA attributable to metastatic disease. Unable to Evaluate (UE): Assigned if bone scan results cannot be interpreted due to inconsistent image acquisition parameters compared to the reference scan, incomplete imaging, or other similar technical deficiencies.
Time Frame: At 24 weeks
Population: Imaging endpt analysis set (IMG): consists of mITT subj. (ITT subj. who received at least one dose of each study drug as randomized) with evaluable imaging scan at baseline, eg. bl quantitated technetium-99 bone scan imaging of sufficient completeness and quality to be assessable and having a non-zero BSLA, as determ. by the central reviewer.
Measure: Number; unit: Percentage
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Radium-223 With Abiraterone & Prednision | Radium-223 With Enzalutamide
Number analyzed (Participants) | 18 | 19 | 16
Percentage
  Responder (R) | 22.2 [10.1 to 39.6] | 57.9 [40.8 to 73.7] | 50.0 [31.8 to 68.2]
  Stable Disease (SD) | 0 | 21.1 | 18.8
  Progressive Disease (PD) | 27.8 | 5.3 | 12.5
  Missing | 50.0 | 15.8 | 18.8
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223); H0: Patient bone scan response rate at Week 24 ≤5%. The Type I error rate for the test in each treatment group, is one-sided 0.10. A one-sided p-value will be reported for this test; Test type: Superiority; p = 0.0109, Clopper and Pearson — [80% CI]: [10.1%- 39.6%]; Patient bone scan response rate at Week 24 will be estimated with exact binomial 80% CI using the method of Clopper and Pearson
Statistical Analysis 2: Comparison: Radium-223 With Abiraterone & Prednision; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Clopper and Pearson — [80% CI]: [40.8% - 73.7%]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Radium-223 With Enzalutamide; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Clopper and Pearson — [80% CI]: [31.8% - 68.2%]; [statistical method as in outcome 1, analysis 1]

2. Primary Outcome: Bone Scan Lesion Area
Description: Bone scan lesion area was defined as the sum of the pixel areas (cm2) of the set of the whole body technetium-99 bone scan imaging pixels identified as bone lesion.
Time Frame: At 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Radium-223 With Abiraterone & Prednision | Radium-223 With Enzalutamide
Number analyzed (Participants) | 18 | 19 | 16
cm^2 | 30227.13 (64912.24) | 10185.58 (12407.65) | 17321.45 (22577.59)

3. Secondary Outcome: Radiological Progression Free Survival
Time Frame: From randomization to radiological disease progression or death from any cause (about 30.82 months )
Population: MITT analysis set: Included all ITT subjects who received at least one dose of each study drug as randomized.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Radium-223 With Abiraterone & Prednision | Radium-223 With Enzalutamide
Number analyzed (Participants) | 19 | 22 | 22
Months | 4.40 [3.75 to 11.5] | NA [18.5 to NA] — NA = Value cannot be estimated due to censored data. | NA [10.15 to NA] — NA = Value cannot be estimated due to censored data.

4. Secondary Outcome: Time to Radiological Progression
Time Frame: From the randomization date to the date of radiological disease progression (about 30.82months)
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Radium-223 With Abiraterone & Prednision | Radium-223 With Enzalutamide
Number analyzed (Participants) | 19 | 22 | 22
Months | 4.40 [3.75 to 11.50] | NA [18.50 to NA] — NA = Value cannot be estimated due to censored data | NA [10.15 to NA] — NA = Value cannot be estimated due to censored data

5. Secondary Outcome: Time to Radiological Bone Progression
Time Frame: From the randomization date to the date of radiological bone progression (about 30.82 months)
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Radium-223 With Abiraterone & Prednision | Radium-223 With Enzalutamide
Number analyzed (Participants) | 19 | 22 | 22
Months | 11.5 [4.40 to 11.5] | NA [NA to NA] — NA = Value cannot be estimated due to censored data | NA [NA to NA] — NA = Value cannot be estimated due to censored data

6. Secondary Outcome: Time to First Symptomatic Skeletal Event
Time Frame: From the randomization date to the first SSE on or following the randomization date (about 30.82 months)
Population: MITT analysis set: Included all ITT subjects who received at least one dose of each study drug as randomized.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Radium-223 With Abiraterone & Prednision | Radium-223 With Enzalutamide
Number analyzed (Participants) | 19 | 22 | 22
Months | NA [12.78 to NA] — NA = Value cannot be estimated due to censored data | NA [17.28 to NA] — NA = Value cannot be estimated due to censored data | NA [19.91 to NA] — NA = Value cannot be estimated due to censored data

7. Secondary Outcome: Symptomatic Skeletal Event-free Survival
Time Frame: From the randomization date to the first SSE on or following the randomization date or death, whichever occurred first (about 32.39 months)
Population: MITT analysis set: Included all ITT subjects who received at least one dose of each study drug as randomized.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Radium-223 With Abiraterone & Prednision | Radium-223 With Enzalutamide
Number analyzed (Participants) | 19 | 22 | 22
Months | 11.93 [10.05 to 24.61] | NA [17.28 to NA] — NA = Value cannot be estimated due to censored data | 19.91 [12.22 to 28.09]

8. Secondary Outcome: Overall Survival
Time Frame: From the randomization date to the date of death due to any cause (about 42.94 months)
Population: MITT analysis set: Included all ITT subjects who received at least one dose of each study drug as randomized.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Radium-223 With Abiraterone & Prednision | Radium-223 With Enzalutamide
Number analyzed (Participants) | 19 | 22 | 22
Months | 35.81 [21.26 to 41.40] | 37.55 [35.88 to NA] — NA = Value cannot be estimated due to censored data | 29.86 [26.58 to NA] — NA = Value cannot be estimated due to censored data

ADVERSE EVENTS:
Time Frame: All AEs occurring from the time the subject signs the ICF until 30 days after the last dose of any study medication (about 18 months).
Groups:
- Radium-223: Radium-223
- Radium-223 + Abiraterone Acetate + Prednisone: Radium-223 + Abiraterone Acetate + Prednisone
- Radium-223 + Enzalutamide: Radium-223 + Enzalutamide
Arm/Group | Radium-223 | Radium-223 + Abiraterone Acetate + Prednisone | Radium-223 + Enzalutamide
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/22 | 1/22
Serious Adverse Events (participants affected / at risk) | 2/19 | 10/22 | 8/22
Other Adverse Events (participants affected / at risk) | 18/19 | 22/22 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 (N=19) | Radium-223 + Abiraterone Acetate + Prednisone (N=22) | Radium-223 + Enzalutamide (N=22)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (8) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (8) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 (N=19) | Radium-223 + Abiraterone Acetate + Prednisone (N=22) | Radium-223 + Enzalutamide (N=22)
Anaemia (Blood and lymphatic system disorders) | 3 (7) | 3 (5) | 3 (5)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 5 (7) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (7) | 8 (15) | 8 (12)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (4) | 9 (11) | 5 (5)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (5) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 3 (3)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 1 (1) | 2 (2) | 1 (1)
Cyst (General disorders) | 0 (0) | 0 (0) | 1 (3)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (9) | 5 (7) | 8 (10)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 3 (4) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 2 (2)
Early satiety (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 4 (4)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (5) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (4)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 1 (2)
Weight decreased (Investigations) | 3 (3) | 1 (1) | 3 (3)
Weight increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (3) | 4 (4) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 3 (6) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 5 (9) | 9 (12)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 3 (3)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 6 (8)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2) | 4 (6)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Apathy (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Middle insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (2)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 2 (2)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (3) | 4 (7)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Systolic hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 3 (3) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 3 (7) | 4 (6) | 4 (6)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 2 (3) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 6 (8) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (7) | 8 (16) | 9 (14)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (4) | 9 (12) | 6 (6)
Vomiting (Gastrointestinal disorders) | 2 (2) | 6 (6) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 3 (3)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 1 (1) | 2 (2) | 1 (1)
Fatigue (General disorders) | 6 (9) | 8 (11) | 9 (11)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 4 (5) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4) | 2 (2)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 5 (5) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 3 (5) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 4 (4)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (5) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 2 (3)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 3 (4) | 1 (3)
Weight decreased (Investigations) | 3 (3) | 1 (1) | 3 (3)
Weight increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (3) | 4 (4) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 3 (6) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (8) | 6 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 8 (13) | 9 (17)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (7) | 4 (6)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 6 (8)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2) | 4 (6)
Headache (Nervous system disorders) | 1 (1) | 5 (5) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 1 (1) | 2 (3)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 3 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 2 (2)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 2 (6) | 6 (13)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days